CLINICAL TRIAL: NCT03459430
Title: The Effect of Core Stability Programs With Different Training Intensities Quantified Using Accelerometers Integrated in Smartphones: a Randomized Controlled Trial
Brief Title: Chronic Effect of Individualized Core Stability Programs in Recreational Athletes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CASTO JUAN RECIO (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government)
Responsible Party: Sponsor-Investigator, CASTO JUAN RECIO, Study Director, Universidad Miguel Hernandez de Elche
Organization: Universidad Miguel Hernandez de Elche (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015/00116/001
Record Dates: First submitted 2018-02-19; First posted 2018-03-08 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Core Stability
Keywords: trunk stability; accelerometer; smartphone; core training; isometric exercises

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low Intensity training group (Experimental): Low Intensity training group will complete a 6 week core stability training program with low intensity/oscillation exercises
  Interventions: Other: Core stability training
- High Intensity training group (Experimental): High Intensity training group will complete a 6 week core stability training program with high intensity/oscillation exercises
  Interventions: Other: Core stability training
- Control group (No Intervention): Control group will have 6 weeks with no intervention before post-test

INTERVENTIONS:
Other: Core stability training — Effect of different core stability programs using diverse training intensities
  Arms: High Intensity training group; Low Intensity training group

SUMMARY:
Core stability (CS) training is nowadays largely used in several fields, mainly to enhance athletic performance and to prevent and rehabilitate musculoskeletal injuries. However, in several experimental studies, CS training programs have not delivered as positive results as could be expected. The lack of proper modulation and quantification of the training load parameters (such as intensity, volume, frequency, etc.) may be one of the main explanations. Although training intensity has been manipulated by modifying the CS exercise difficulty through variations in mechanical constraints (i.e. participant posture, lever arms, base of support, unstable surfaces, etc.), to the best of the authors' knowledge no experimental study has quantified the CS training intensity based on objective parameters. The quantification of the load intensity is fundamental to analyze the dose-response relationships between training and CS adaptations. Therefore, the main aim of this study is to evaluate the effectiveness of two individualized CS training programs using smartphone accelerometers placed on the pelvis to quantify the intensity of several of the most common CS exercises employed in fitness, sports and rehabilitation. The expected effect is that the experimental groups will improve CS significantly.

DETAILED DESCRIPTION:
Sixty recreational male athletes will be evaluated twice (pre-test 1 and pre-test 2) before a core stability (CS) training program. Testing sessions will consist in several tests to assess sitting and global dynamic postural control, trunk isometric endurance, neuromuscular function of the lower extremities, trunk response to sudden and unexpected load perturbations and pelvic oscillation during CS exercises evaluated with a smartphone accelerometer. Later, they will be randomly assigned to one of the three groups included in the study: two experimental groups (low and high intensity) and a control group. The intervention will have a training frequency of 2 days per week for 6 weeks. Each CS training session will consist in 4 sets of one variation of four of the most popular stabilization exercises used to challenge core muscles: frontal bridge, back bridge, lateral bridge and bird-dog. Exercise variations will be performed isometrically in increasing order of difficulty through the modifications of the following mechanical constraints: lever-arm, number of supports and/or the use of unstable surfaces. The CS training programs will differ in exercises intensity, mainly. Each participant of the low intensity group will perform those exercise variations in which they have obtained an oscillation ranged between 0.2 and 0.3 m/s2 in pre-test, while participants of the high intensity group will perform the exercise variations in which they have obtained an oscillation ranged between 0.4 and 0.5 m/s2. The exercise duration will be set at 30 s and 15 s for the low intensity and high intensity group, respectively. All participants of the training groups will be revaluated every two weeks during the training period. After the intervention period, all participants will perform a post-test to evaluate the effectiveness of both CS programs. Statistical analysis will consist in repeated-measures ANOVAs for detecting possible significant differences within and between-groups.

ELIGIBILITY:
Inclusion Criteria:

- Healthy recreative male athletes between 18 and 35 years old

Exclusion Criteria:

* Inguinal hernia or urinary incontinence
* Pathologies that contraindicate physical exercise practice
* Low back pain in the last six months prior to testing
* Pathologies related with Central Nervous System that affect balance
* Professional athletes of sports modalities with high core stability demands

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-03-10 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
Mean radial error of center of pressure in sitting condition | Baseline - 6 weeks
  Postural control in sitting condition over an unstable seat evaluated through the mean radial error of center of pressure displacement (Units: millimeters)
Trunk angular displacement | Baseline - 6 weeks
  Trunk angular displacement after sudden loading perturbations in different planes of motion (units: degrees)
Pelvis mean acceleration | Baseline - every 2 weeks up to 6 weeks
  Pelvis mean acceleration in different isometric stabilization exercises measured with a smartphone accelerometer (Units: m/s2)

OTHER OUTCOMES:
Global dynamic balance in anterior direction | Baseline - 6 weeks
  Anterior reaching distance during unipodal stance (units: centimeters)
Global dynamic balance in posteromedial direction | Baseline - 6 weeks
  Posteromedial reaching distance during unipodal stance (units: centimeters)
Global dynamic balance in posterolateral direction | Baseline - 6 weeks
  Posterolateral reaching distance during unipodal stance (units: centimeters)
Mean radial error of center of pressure in upright tandem stance | Baseline - 6 weeks
  Postural control in upright tandem stance condition evaluated through the mean radial error of center of pressure displacement (Units: millimeters)
Trunk extensors isometric endurance | Baseline - 6 weeks
  Time to maintain a particular position against gravity until exhaustion using Biering-Sorensen test; (Units: seconds)
Trunk flexors isometric endurance | Baseline - 6 weeks
  Time to maintain a particular position against gravity until exhaustion using using Plank test; (Units: seconds)
Trunk lateral flexors isometric endurance | Baseline - 6 weeks
  Time to maintain a particular position against gravity until exhaustion using Side Bridge test; (Units: seconds)
Neuromuscular function of lower extremity | Baseline - 6 weeks
  Triple hop test (Units: centimeters)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco J Vera-Garcia, Professor, Principal Investigator — Universidad Miguel Hernandez de Elche, Spain
Locations (1):
- Sport Research Center, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Yes
All Individual Participant Data (IPD) that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available six months after publication
Access Criteria: Data access requests will be reviewed by an external Independent Review Panel. Requestors will be required to sign a Data Access Agreement